CLINICAL TRIAL: NCT03512535
Title: Method Validation for New Nitrogen/Sulfur Species Analysis Techniques
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Southampton (Other)
Responsible Party: Sponsor
Other Study IDs: 31426
Record Dates: First submitted 2018-04-18; First posted 2018-04-30 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Redox Status

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, serum and whole blood pellets
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stage 1: Samples from up to 20 participants will be used to finalise the analytical methods
- Stage 2: Samples from up to 200 participants will be used to then validate the normal ranges of these markers across different age ranges in both genders

SUMMARY:
Plasma redox status is well known to alter with age but previously differences have only been reported for two specific redox couples; reduced and oxidized cysteine and reduced and oxidized glutathione. (Jones DP, Rejuvenation Res. 2006) The overall aim of this project is to develop new methods to determine how other Reactive Nitrogen and Sulfur species, such as free and protein-bound thiols (organic compounds that contain a Sulfhydryl group, -SH) and Hydrogen Sulfide (H2S) change with age and gender in a medium-sized cohort of healthy individuals (n=100 of either sex; age 18-70).

Our group has recently developed a novel analytical platform to measure thiol-containing compounds in biological samples that is based on the reaction with the thiol-alkylating agent N-ethylmaleimide (NEM). We have used this chemical for years as stabilisation agent in other analyses to quantify Nitric Oxide metabolites.(Feelisch et al, FASEB 2002 and Levett et al, Sci Rep 2011) We now wish to develop a similar method to measure thiol containing compounds using a novel rapid LC-MS/MS based technology for screening large numbers of individuals.

The project will therefore have 2 stages:

1. Initial method development will require occasional use of whole blood, plasma and red blood cells to establishing optimal conditions. E.g. to compare heparin and EDTA as anticoagulants to serum; investigate effects of temperature and pH; identify optimal concentration of derivatisation/reduction agents and optimal reaction times.
2. We then aim to establish the normal distribution of these novel compounds across healthy individuals of different gender and varying ages.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or above
* Currently healthy (i.e. no inter-current illness/infection)
* Capacity and ability to give written informed consent

Exclusion Criteria:

* Current or previous smoker
* Other medical co-morbidity (e.g. hypertension, diabetes, asthma, COPD, cardiovascular disease, current or previous malignant disease etc.)
* Surgery within previous 28 days
* Excessive alcohol intake (i.e above UK's recommended intake limit of 14 units per week).
* Pregnant or currently breast-feeding
* On current medication
* Taken vitamins / minerals / herbal remedies within previous 28 days
* Difficult venous access
* Needle phobia
* Participating in another similar/conflicting research study already

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy adult volunteers
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2018-01-29 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Concentration of reactive (nitrogen or sulfur containing) species | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Martin Feelisch, PhD, Study Chair — University of Southampton
Locations (1):
- University of Southampton, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided